CLINICAL TRIAL: NCT07159126
Title: A Phase 1, Open-label, Multicenter, First-in-Human Trial of DS3610a in Participants With Advanced Solid Tumor
Brief Title: A Study of DS3610a in Participants With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3610-071; 2025-521173-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors; Metastatic Solid Tumors
Keywords: DS3610a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS3610a at Escalating Doses (Experimental): Participants will receive DS3610a at escalating doses.
  The RDE will be determined using data collected from this arm.
  Interventions: Drug: DS3610a

INTERVENTIONS:
Drug: DS3610a — Participants will receive DS3610a at the target dose. Treatment will continue until radiographic disease progression, as determined by the investigator, or until another reason for discontinuation of trial intervention occurs.

SUMMARY:
This study is designed to assess the safety, tolerability, and efficacy of DS3610a, given as a single agent to participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a dose escalation study for participants with advanced or metastatic solid tumors. The primary objective of the study is to determine the Recommended Dose for Expansion (RDE), and to evaluate the safety, tolerability, PK, and preliminary efficacy of DS3610a in solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Sign and date the main ICF, prior to the start of any trial-specific procedures.
* Adults ≥18 years of age at the time the ICF is signed (Please follow local regulatory requirements if the legal age of consent for trial participation is >18 years old).
* Relapsed from, refractory to, or intolerant to appropriate therapies (eg, SoC) to provide clinical benefit for their condition as assessed by their physician and/or investigator.
* Is willing and able to provide an adequate pretreatment tissue sample prior to trial intervention or archival tumor tissue sample.
* Has measurable disease based on local CT/MRI imaging as assessed by the investigator per RECIST v1.1; radiographic tumor assessment must be performed within 28 days prior to initiation of trial intervention.

Key Exclusion Criteria:

*Inadequate washout period before initiation of trial intervention, defined as: Major surgery: ≤4 weeks (or ≤2 weeks for low-invasive cases) Curative radiation therapy: ≤4 weeks Chemotherapy, Ab-based anticancer therapy, immunotherapy: ≤4 weeks Small molecules (eg, tyrosine kinase inhibitors): ≤2 weeks or 5 half-lives, whichever is longer Nitrosoureas: ≤6 weeks

* Has known symptomatic CNS metastases, leptomeningeal disease, or cord compression. Note: Asymptomatic or adequately treated CNS metastases are not exclusionary provided that, in the opinion of the investigator, the participant is neurologically stable. MRI/CT of the brain is required for all participants during SCR Period
* Uncontrolled or clinically significant cardiovascular disease, including the following:

  1. Myocardial infarction within 6 months prior to SCR.
  2. Uncontrolled angina pectoris within 6 months prior to SCR.
  3. New York Heart Association (NYHA) Class III or IV CHF.
  4. LVEF ≤50%.
  5. QTcF interval >470 ms.
* Any of the following within the past 6 months prior to enrollment: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic events.
* Clinically severe pulmonary compromise (ie, requiring any supplemental oxygen) resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the trial enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion, etc.) and any autoimmune, connective tissue, or inflammatory disorder with potential pulmonary involvement (eg, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or prior pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | From first dose, up to approximately 24 months

SECONDARY OUTCOMES:
Area Under the Blood Concentration-time Curve During Dosing Interval | From baseline to postbaseline, up to approximately 36 months
  Area Under the Blood Concentration-time Curve During Dosing Interval (AUCtau) will be used to asses PK parameters
Antidrug Antibody Prevalence | From baseline to postbaseline, up to approximately 36 months
  The percentage of participants who are Antidrug Antibody positive at any point in time.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/